CLINICAL TRIAL: NCT02048215
Title: Evaluation of Diet and Treatment With a Combination of Ephedrine and Caffeine on Thermogenesis, Cardiac Function and on Uncoupling Proteins Expression in Adipose and Muscle Tissue of Morbid Obese Patients Undergoing Bariatric Surgery.
Brief Title: Effect on Energy Metabolism at Cellular Level of Diet Plus Treatment With Ephedrine and Caffeine in Obesity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: University of Milan (Other); Università Politecnica delle Marche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: THERMODIET
Record Dates: First submitted 2014-01-22; First posted 2014-01-29 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Obesity
Keywords: thermogenesis; low-calorie diet; uncoupling-protein 3; beta-3 adrenoceptors; thermogenic drugs
MeSH Terms: conditions — Obesity | interventions — Caffeine; Ephedrine; Caloric Restriction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ephedrine + Caffeine + diet (Active Comparator): Ephedrine 20 mg + Caffeine 200 mg capsule t.i.d. for one month plus hypocaloric diet
  Interventions: Drug: Caffeine; Drug: Ephedrine; Other: Hypocaloric diet
- Placebo + diet (Placebo Comparator): Similarly-looking placebo capsule t.i.d. for one month plus hypocaloric diet
  Interventions: Drug: Placebo; Other: Hypocaloric diet

INTERVENTIONS:
Drug: Caffeine — Patients are randomised to 30-day treatment with either EC (200/20mg t.i.d.) or placebo. The EC administration starts with an initial dose of 100/10 mg t.i.d. for the first week and then proceeds with the full dose of 200/20 mg t.i.d. Patients are hospitalised during the whole treatment period, at the metabolic unit of San Giuseppe Hospital-Istituto Auxologico Italiano at Piancavallo (VB, Italy). During the treatment period all patients are fed a hypocaloric diet (total energy content of ~70% of energy expenditure, as measured by indirect calorimetry), and containing 20% proteins, 55% carbohydrates, 25% fat half of which was monounsaturated, and 35 g/day fibres.
  Other Names: Randomization number 2, 4, 5, 6, 8, 11
  Arms: Ephedrine + Caffeine + diet
Drug: Placebo — Patients are randomised to 30-day treatment with either EC (200/20mg t.i.d.) or placebo. The EC administration starts with an initial dose of 100/10 mg t.i.d. for the first week and then proceeds with the full dose of 200/20 mg t.i.d. Patients are hospitalised during the whole treatment period, at the metabolic unit of San Giuseppe Hospital-Istituto Auxologico Italiano at Piancavallo (VB, Italy). During the treatment period all patients are fed a hypocaloric diet (total energy content of ~70% of energy expenditure, as measured by indirect calorimetry), and containing 20% proteins, 55% carbohydrates, 25% fat half of which was monounsaturated, and 35 g/day fibres.
  Other Names: Randomization number 1, 3, 7, 9, 10, 12, 13
  Arms: Placebo + diet
Drug: Ephedrine — Patients are randomised to 30-day treatment with either EC (200/20mg t.i.d.) or placebo. The EC administration starts with an initial dose of 100/10 mg t.i.d. for the first week and then proceeds with the full dose of 200/20 mg t.i.d. Patients are hospitalised during the whole treatment period, at the metabolic unit of San Giuseppe Hospital-Istituto Auxologico Italiano at Piancavallo (VB, Italy). During the treatment period all patients are fed a hypocaloric diet (total energy content of ~70% of energy expenditure, as measured by indirect calorimetry), and containing 20% proteins, 55% carbohydrates, 25% fat half of which was monounsaturated, and 35 g/day fibres.
  Other Names: Randomization number 2, 4, 5, 6, 8, 11
  Arms: Ephedrine + Caffeine + diet
Other: Hypocaloric diet — Patients are randomised to 30-day treatment with either EC (200/20mg t.i.d.) or placebo. The EC administration starts with an initial dose of 100/10 mg t.i.d. for the first week and then proceeds with the full dose of 200/20 mg t.i.d. Patients are hospitalised during the whole treatment period, at the metabolic unit of San Giuseppe Hospital-Istituto Auxologico Italiano at Piancavallo (VB, Italy). During the treatment period all patients are fed a hypocaloric diet (total energy content of ~70% of energy expenditure, as measured by indirect calorimetry), and containing 20% proteins, 55% carbohydrates, 25% fat half of which was monounsaturated, and 35 g/day fibres.
  Other Names: Low-calorie diet 70% of measured energy expenditure

SUMMARY:
Brief Summary This trial was part of a sub-project targeted to diet, thermogenesis and obesity of a larger multicentre study named "Interaction between nutritional, social-behavioral and metabolic factors for prevention of cardiovascular disease: development of nutritional strategies on general population".

Ephedrine and caffeine (EC) combination has been widely used in human obesity treatment. It is known that this drug increases the metabolic rate in both animals and humans. Ephedrine is an agonist of both α and β-adrenoceptors; moreover, it induces norepinephrine release from sympathetic neurons. Caffeine increases both norepinephrine and dopamine release and stimulates the neuronal activity in several brain regions. We hypothesize that EC treatment might exert a specific effect on lipolysis and thermogenesis by stimulation of beta-3 adrenoreceptors on adipose tissue and by stimulating uncoupling of oxidative phosphorylation, i.e. energy being dissipated as heat rather than being converted to adenosine triphosphate (ATP)

Our study is a double-blind, placebo-controlled, 4-week trial to investigate the effect of hypocaloric diet alone or coupled to EC treatment of morbidly obese women on thermogenesis, expression of UCP 3 (in muscle tissue) and of beta-3 adrenoreceptors (in adipose tissue). Subjects are randomly assigned to EC (200/20 mg) or to placebo administered three times a day orally together with a energy-deficit diet (70% of resting energy expenditure), starting one month before undergoing bariatric surgery. Primary study endpoints are weight change analysed by intention to treat, changes in resting energy expenditure, UCP3 (long and short isoform), messenger ribonucleic acid (mRNA) levels in rectus abdominis and immunostaining for beta-3 adrenoreceptors in subcutaneous and omental adipose tissue. Also plasma epinephrine, norepinephrine, triglycerides, free fatty acids, glycerol, TSH, free thyroxine (fT4), free triiodothyronine (fT3) fasting glucose, insulin and homeostasis model assessment (HOMA) index, are measured at baseline and at the end of treatments.

DETAILED DESCRIPTION:
This trial was part of a sub-project of a multicentre study named "Interaction between nutritional, social-behavioral and metabolic factors for prevention of cardiovascular disease: development of nutritional strategies on general population" approved by the Italian Ministry of Health. The sub-project was specifically addressed to diet, thermogenesis and obesity.

1. Ephedrine and caffeine (EC) combination has been widely used in human obesity treatment, and is still present in many herbal preparations sold widespread in many countries for weight loss. It is well known that this drug increases the metabolic rate in both animals and humans. Ephedrine is an agonist of both α and β-adrenoceptors; moreover, it induces norepinephrine release from sympathetic neurons, and thus is a sympatho-mimetic drug with a mixed profile. Caffeine increases both norepinephrine and dopamine release and stimulates the neuronal activity in several brain regions. In addition, caffeine antagonizes the inhibitory effects of adenosine on sympathetic nervous system (SNS). This modulation of SNS activity may be a possible explanation for the thermic effect of EC. In fact, epinephrine activates the uncoupling protein 1 (UCP1), a member of mitochondrial carriers localized on the inner mitochondrial membrane in brown adipocytes. The physiological role of UCP1 is to uncouple oxidative phosphorylation, therefore most of the energy is dissipated as heat rather than being converted to ATP. UCP1 is unique to brown adipocyte mitochondria, although brown-like multilocular adipocytes expressing UCP1 interspersed within human WAT have been observed. Actually, UCP1 mRNA has been detected in all adipose tissues in adult humans, and it has been estimated that 1 in 100-200 adipocytes in human intraperitoneal adipose tissue expresses UCP1. It has been shown that the cold-induced occurrence of brown-like adipocytes and UCP1 requires the presence of the β3-adrenoceptor in previously white adipose tissue and the presence of the β3-adrenoceptor is required for full stimulation of energy expenditure and oxygen consumption in white adipose tissue.

   In addition to UCP1, expressed exclusively in brown adipose tissue (BAT), another member of the mitochondrial anion carrier protein family i.e. uncoupling protein 3 (UCP3) could play a physiological role in energy homeostasis. It is expressed almost exclusively in skeletal muscle and exhibits two transcriptional isoforms: a long form (UCP3L) and a short form (UCP3S). A brief caloric restriction resulted in ~2- to 3-fold increase in UCP3 mRNA levels in lean and obese humans.
2. Because only a few, small studies have been done in humans to investigate the thermogenic effects of EC as compared to diet only, in the present study we examined the UCP3 expression in skeletal muscle and the beta-3 adrenoceptor expression in adipose tissue of pre-menopausal morbidly obese females treated with either placebo or EC for 30 days who subsequently underwent bariatric surgery.
3. Study subjects are adult females with morbid obesity i.e. body mass index ≥ 40 kg/m2 selected from the waiting list for bariatric surgery at Department of Surgery (Molinette Hospital, Turin, Italy. During the treatment period all patients are fed a hypocaloric diet (total energy content of ~70% of energy expenditure, as measured by indirect calorimetry), and containing 20% proteins, 55% carbohydrates, 25% fat half of which was monounsaturated, and 35 g/day fibres. Patients are randomised to 30-day treatment with either EC (200/20mg t.i.d.) or placebo. They are hospitalised, during the whole treatment period, at the metabolic unit of San Giuseppe Hospital-Istituto Auxologico Italiano at Piancavallo (VB, Italy). The EC administration starts with an initial dose of 100/10 mg t.i.d. for the first week and then proceeds with the full dose of 200/20 mg t.i.d. Resting energy expenditure is measured by indirect calorimetry at baseline and at the end of the study. The study pills (active compound and placebo) were prepared by the Hospital's Pharmacy.
4. In order to evaluate drug safety and effect on cardiac function, the blood pressure is measured three times a day; both electrocardiography and echocardiography are being recorded at baseline and every week. After diet and drug period, the patients are transferred to the Department of Surgery (Molinette Hospital, Turin) for the bariatric surgery. The drug treatment (EC and placebo) is stopped the day before surgical intervention. Small biopsies of rectus abdominis and of subcutaneous and omental adipose tissues are taken during surgery, immediately frozen in liquid nitrogen, and stored at -80°C for subsequent analysis.
5. UCP3S and UCP3L mRNA levels are measured by quantitative polymerase chain reaction at the Department of Pharmacology, University of Milan. Presence of beta-3 adrenoceptor in adipose tissue is evaluated by immunohistochemistry by the avidin-biotin peroxidase technique using monoclonal anti-human beta 3-adrenoceptor antibody at the Department of Human Anatomy, University of Ancona.

ELIGIBILITY:
Inclusion Criteria:

* pre-menopausal females
* body mass index ≥ 40 kg/m2
* with stable weight in the three month before the study
* scheduled for bariatric surgery
* in whom weight loss was clinically advisable before surgery to reduce surgical risk
* non-smokers or smoking less than 5 cigarettes per day

Exclusion Criteria:

* pregnancy
* ischaemic heart disease
* cardiac failure
* high blood pressure requiring drug treatment
* tachyarrhythmia
* sick sinus syndrome
* atrioventricular block
* two-bundle ventricular block
* cerebrovascular diseases
* occlusive peripheral artery disease
* renal failure
* current treatment with drugs that might affect metabolic rate (e.g. β-adrenergic blockers, thyroid hormones).

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2000-02; Primary Completion 2001-01 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Change in resting energy expenditure | Baseline and 1 month
  Resting energy expenditure is measured by indirect calorimetry

SECONDARY OUTCOMES:
Blood pressure monitoring | Baseline and daily for 30 days (t.i.d.)
Electrocardiograpic monitoring | Baseline and at week 2,3,4
Cardiac ultrasound monitoring | Baseline and at week 2,3,4
  Cardiac ultrasound measurement for assessing possible detrimental changes
Changes in fasting glucose | Baseline and at one month
  Patients are assessed by oral glucose tolerance test at baseline and following one month of treatment, with assessment of glucose, insulin, free-fatty acids and glycerol
Changes in fasting insulin | baseline and one month
  Patients are assessed by oral glucose tolerance test at baseline and following one month of treatment, with assessment of glucose, insulin, free-fatty acids and glycerol
Changes in fasting free fatty acids | baseline ans one month
  Patients are assessed by oral glucose tolerance test at baseline and following one month of treatment, with assessment of glucose, insulin, free-fatty acids and glycerol
Changes in fasting glycerol | baseine and one month
  Patients are assessed by oral glucose tolerance test at baseline and following one month of treatment, with assessment of glucose, insulin, free-fatty acids and glycerol
Changes in thyroid function (TSH, T3, T4) | Baseline and 1 month
Changes in plasma noradrenalin | Baseline and 1 month
Changes in body weight | baseline and 1 month
Beta-3 adrenoceptor expression in human adipose tissue | one month
  Beta-3 adrenoceptor expression is measured in subcutaneous and omental tissue sampled during bariatric surgery following one month of pharmacological intervention
UCP-3 expression in human muscle tissue | One month
  UCP-3 expression is measured in rectus abdominis muscle tissue sampled during bariatric surgery following one month of pharmacological intervention

CONTACTS AND LOCATIONS:
Overall Officials: Maria L Petroni, MD, Principal Investigator — Istituto Auxologico Italiano
Locations (1):
- Istituto Auxologico Italiano -Ospedale San Giuseppe, Verbania, VB, Italy

REFERENCES:
- [Background] Dulloo AG, Miller DS. The thermogenic properties of ephedrine/methylxanthine mixtures: human studies. Int J Obes. 1986;10(6):467-81. PMID 3804564
- [Background] Astrup A, Breum L, Toubro S. Pharmacological and clinical studies of ephedrine and other thermogenic agonists. Obes Res. 1995 Nov;3 Suppl 4:537S-540S. doi: 10.1002/j.1550-8528.1995.tb00224.x. PMID 8697055
- [Background] Miller DS, Stock MJ, Stuart JA. Proceedings: The effects of caffeine and carnitine on the oxygen consumption of fed and fasted subjects. Proc Nutr Soc. 1974 Sep;33(2):28A-29A. No abstract available. PMID 4456386
- [Background] Acheson KJ, Zahorska-Markiewicz B, Pittet P, Anantharaman K, Jequier E. Caffeine and coffee: their influence on metabolic rate and substrate utilization in normal weight and obese individuals. Am J Clin Nutr. 1980 May;33(5):989-97. doi: 10.1093/ajcn/33.5.989. PMID 7369170
- [Background] Astrup A, Toubro S, Christensen NJ, Quaade F. Pharmacology of thermogenic drugs. Am J Clin Nutr. 1992 Jan;55(1 Suppl):246S-248S. doi: 10.1093/ajcn/55.1.246s. PMID 1345887
- [Background] Bellet S, Roman L, DeCastro O, Kim KE, Kershbaum A. Effect of coffee ingestion on catecholamine release. Metabolism. 1969 Apr;18(4):288-91. doi: 10.1016/0026-0495(69)90049-3. No abstract available. PMID 5777013
- [Background] Berkowitz BA, Spector S. Effect of caffeine and theophylline on peripheral catecholamines. Eur J Pharmacol. 1971 Jan;13(2):193-6. doi: 10.1016/0014-2999(71)90150-6. No abstract available. PMID 5544072
- [Background] Klaus S, Casteilla L, Bouillaud F, Ricquier D. The uncoupling protein UCP: a membraneous mitochondrial ion carrier exclusively expressed in brown adipose tissue. Int J Biochem. 1991;23(9):791-801. doi: 10.1016/0020-711x(91)90062-r. No abstract available. PMID 1773883
- [Background] Garruti G, Ricquier D. Analysis of uncoupling protein and its mRNA in adipose tissue deposits of adult humans. Int J Obes Relat Metab Disord. 1992 May;16(5):383-90. PMID 1319974
- [Background] Lean ME, James WP, Jennings G, Trayhurn P. Brown adipose tissue in patients with phaeochromocytoma. Int J Obes. 1986;10(3):219-27. PMID 3019909
- [Background] Oberkofler H, Dallinger G, Liu YM, Hell E, Krempler F, Patsch W. Uncoupling protein gene: quantification of expression levels in adipose tissues of obese and non-obese humans. J Lipid Res. 1997 Oct;38(10):2125-33. PMID 9374134
- [Background] Grujic D, Susulic VS, Harper ME, Himms-Hagen J, Cunningham BA, Corkey BE, Lowell BB. Beta3-adrenergic receptors on white and brown adipocytes mediate beta3-selective agonist-induced effects on energy expenditure, insulin secretion, and food intake. A study using transgenic and gene knockout mice. J Biol Chem. 1997 Jul 11;272(28):17686-93. doi: 10.1074/jbc.272.28.17686. PMID 9211919
- [Background] Solanes G, Vidal-Puig A, Grujic D, Flier JS, Lowell BB. The human uncoupling protein-3 gene. Genomic structure, chromosomal localization, and genetic basis for short and long form transcripts. J Biol Chem. 1997 Oct 10;272(41):25433-6. doi: 10.1074/jbc.272.41.25433. PMID 9325252
- [Background] Millet L, Vidal H, Andreelli F, Larrouy D, Riou JP, Ricquier D, Laville M, Langin D. Increased uncoupling protein-2 and -3 mRNA expression during fasting in obese and lean humans. J Clin Invest. 1997 Dec 1;100(11):2665-70. doi: 10.1172/JCI119811. PMID 9389729
- [Result] De Matteis R, Arch JR, Petroni ML, Ferrari D, Cinti S, Stock MJ. Immunohistochemical identification of the beta(3)-adrenoceptor in intact human adipocytes and ventricular myocardium: effect of obesity and treatment with ephedrine and caffeine. Int J Obes Relat Metab Disord. 2002 Nov;26(11):1442-50. doi: 10.1038/sj.ijo.0802148. PMID 12439645
- [Derived] Bracale R, Petroni ML, Davinelli S, Bracale U, Scapagnini G, Carruba MO, Nisoli E. Muscle uncoupling protein 3 expression is unchanged by chronic ephedrine/caffeine treatment: results of a double blind, randomised clinical trial in morbidly obese females. PLoS One. 2014 Jun 6;9(6):e98244. doi: 10.1371/journal.pone.0098244. eCollection 2014. PMID 24905629